CLINICAL TRIAL: NCT06719713
Title: Store Safely: Rural Firearm Injury Prevention for Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Marquette County Health Department (Unknown)
Responsible Party: Principal Investigator, Cynthia Ewell Foster, Clinical Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00250518; 1 R01CE003629-01-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 1R01CE003629-01 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Firearm Injury
Keywords: rural; firearm safe storage; injury prevention; suicide prevention; community education
MeSH Terms: conditions — Suicide Prevention; Health Education

STUDY DESIGN:
Intervention Model Description: Waitlist control and intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Store Safely (Experimental): The Store Safely arm (consisting of a community sample) will receive the Store Safely intervention, usual community-based care, and 988 suicide and crisis lifeline number and a publicly available safe storage information resource numbers.
  Interventions: Behavioral: Store Safely
- Waitlist control (No Intervention): The waitlist control group (consisting of a community sample) will not receive the intervention during the clinical trial but will be offered 988 suicide and crisis lifeline number and a publicly available safe storage information resource numbers. Following the clinical trial they will have access to the Store Safely intervention.

INTERVENTIONS:
Behavioral: Store Safely — The Store Safely intervention occurs online and is self-administered. Once directed to the Store Safely website, participants are welcomed and instructed to complete each step of the online program. Upon clicking "Start," participants are taken to Step 1 of the intervention and instructed to review a brief video. Step 2 involves a review of a data infographics. Participants are then directed to the Decision Aid in Step 3. In Step 4, participants are instructed to complete the Family Firearm Storage Action Plan. In Step 5, participants will review another brief video. There will also be an optional step, consisting of a resource page that details local options for obtaining safe storage devices. At the end of each step, participants mark a checkbox to indicate they have completed the intervention activity which facilitates website analytics of participant engagement. Lastly, participants are thanked and provided with details about the final steps of the trial.
  Arms: Store Safely

SUMMARY:
The researchers are testing a firearm safety prevention strategy tailored for families with children who reside in a rural area. Researchers hypothesize that the intervention will lead to improvements in household firearm storage.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* English-speaking
* Have a child under 18 living at home
* Own at least one firearm
* Reside in Michigan's Upper Peninsula (UP)
* Access to a computer/mobile device and wifi
* Have sufficient information about household storage to complete surveys

Exclusion Criteria:

* Unable to be consented in English
* Lack of firearm in the home
* No child in the home
* Residence outside the UP
* No access to technology
* Previously enrolled in 2020 pilot project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of firearms stored locked | Approximately 3 months
  Measured using a self-report item from the Family Firearm Storage Behaviors Survey (Ewell Foster et al., 2024) administered at 3 months. May range from 1-40 based on pilot data
Parent Engagement in Harm Reduction Firearm Storage Behaviors Score | Approximately 3 months
  Measured using the Family Firearm Storage Behaviors Survey (Ewell Foster et al., 2024) administered at 3 months. The survey is 14 items, endorsed as Y/N. Score range is 0-14.

SECONDARY OUTCOMES:
Parent Self-Efficacy for Firearm Safety Questionnaire | Baseline, Immediate/2-Week
Number of firearms unloaded | Approximately 3 months
  Measured using a self-report item from the Family Firearm Storage Behaviors Survey (Ewell Foster et al., 2024) administered at 3 months.
Number of firearms unlocked and loaded | Approximately 3 months
  Measured using a self-report item from the Family Firearm Storage Behaviors Survey (Ewell Foster et al., 2024) administered at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ewell Foster, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Marquette County Health Department, Negaunee, Michigan

IPD SHARING:
Plan to Share IPD: Yes
After the study is complete and data has been cleaned and de-identified, the archived data will be transmitted to and securely stored at the University of Michigan Institute for Firearm Injury Prevention Data Repository, for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, ICF
Time Frame: After the study is completed and available according to Firearm Injury Prevention Data Repository policy.
Access Criteria: Researchers can request data from the study contacts listed in the study.
URL: https://firearminjury.umich.edu/data-reporting/